CLINICAL TRIAL: NCT04737902
Title: Erector Spinae Plane (ESP) Block, Incidence of Chronic Neuropathic Pain (CNP) and Quality of Life (QoL) After VATS. An Observational Study.
Brief Title: ESP Block, CNP and QoL After VATS
Status: Completed | Type: Observational
Sponsor: Hospital Universitario San Ignacio (Other)
Responsible Party: Sponsor
Other Study IDs: FMCIE-0043-19
Record Dates: First submitted 2021-01-30; First posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-01

CONDITIONS: Postoperative Pain; Video-assisted Thoracoscopic Surgery
Keywords: regional anesthesia; postoperative pain; video-assisted thoracoscopic surgery; erector spinae plane block; Neuropathic Pain; Quality of Life
MeSH Terms: conditions — Pain, Postoperative; Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- VATS with ESPB: Study subjects underwent anaesthesia and VATS without a change in their routine care. At the end of the surgery, an erector spinae plane block was performed for acute pain control following our institutional protocol for perioperative care.
  Interventions: Procedure: Erector spinae plane block

INTERVENTIONS:
Procedure: Erector spinae plane block — Unilateral ESP block was performed between T3 and T7 levels depending on the thoracic surgical incision. The patient is placed in lateral decubitus position, under sterile conditions, a high frequency (6-15 MHz) linear-array transducer (Sonosite® Edge II, Bothell, USA) was placed in a longitudinal parasagittal orientation 2 cm from the posterior midline to visualise the tips of the transverse processes deep to the erector spinae muscle (ESM). A 21 G, 50 mm or 100 mm needle (Pajunk UniPlex NanoLine; Germany) was advanced in-plane with the ultrasound beam. The needle tip was directed to the plane between the transverse process and the posterior fascia of the ESM. Correct needle tip location was confirmed by ultrasound visualisation of linear fluid spread in the fascial plane. The injection of 0.5 to 1 ml of bupivacaine was 0.5% with epinephrine 5 µg/ml; then, a total of 20-30 ml of the same local anaesthetic was administered.

SUMMARY:
The Erector Spinae Plane Block (ESPB) is an adequate alternative for pain management after video-assisted thoracoscopy surgery (VATS). The incidence of postoperative chronic neuropathic pain (CNP) and the quality of life (QoL) in patients with ESPB after VATS remain unknown. We hypothesised that patients with ESPB would have a low incidence of acute and CNP and would report a good QoL up to three months after VATS.

DETAILED DESCRIPTION:
We, therefore, performed this prospective observational study. The a priori primary outcome was incidence of CNP three months postoperatively (POP) in patients undergoing VATS surgery with ESPB as the regional anaesthesia technique. The secondary outcome was to describe pain control at PACU, 12 and 24 hours POP and QoL reported up to three months after surgery. We hypothesised that patients with ESPB would have a low incidence of acute and CNP and report a good QoL.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent VATS and required at least one day of hospital stay after surgery

Exclusion Criteria:

* patients with mental or physical limitation to answer the questionnaires.
* patients who required mechanical ventilation.
* patients who required surgery conversion to thoracotomy.
* patients who declined consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Incidence of chronic neurophatic pain | 3 month
  incidence of CNP three months postoperatively (POP) in patients undergoing VATS surgery with ESPB as the regional anaesthesia technique

SECONDARY OUTCOMES:
Postoperative pain | 24 hours
  pain control at PACU, 12 and 24 hours POP
Quality of Life POP | 3 months POP
  Quality of Life by EQ-5D

CONTACTS AND LOCATIONS:
Overall Officials: Lorena Díaz-Bohada, MD, MSc, Principal Investigator — Hospital Universitario San Ignacio
Locations (1):
- Hospital Universitario, Bogota, Cundinamarca, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bayman EO, Parekh KR, Keech J, Selte A, Brennan TJ. A Prospective Study of Chronic Pain after Thoracic Surgery. Anesthesiology. 2017 May;126(5):938-951. doi: 10.1097/ALN.0000000000001576. PMID 28248713
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016